CLINICAL TRIAL: NCT06790173
Title: Effects of Strategy Training for Physical Activity on Executive Functions in Stroke Survivors With Cognitive Impairments: a Phase II Randomized Controlled Trial
Brief Title: Effects of Strategy Training for Physical Activity (STPA) on the Post-stroke Executive Dysfunction
Acronym: STPA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202405115
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Executive function; Strategy training; Physical activity
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Intervention Model Description: The allocation ratio is 1:1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A researcher is responsible for the randomization process and the results are coded with predefined IDs that investigators and outcomes assessors are unaware of the meaning.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strategy training for physical activity (Experimental): Trained therapists visit each participant for 60 minutes twice or thrice a week. The program consists of 12 therapist-guided sessions over a maximum of 6 weeks and includes the following active ingredients: knowledge of physical activity, self-selected activity-based goals, dynamic performance analysis, global strategy ("Goal-PlanDo-Check"), and guided discovery.
  Interventions: Behavioral: Strategy training for physical activity
- Physical activity (Active Comparator): Participants assigned to the PA group receive a protocol of exercise program with 12, 1-hour sessions in total. Similar to STPA group, the frequency of intervention is twice or thrice a week.
  Interventions: Behavioral: Physical activity
- Education (Active Comparator): Participants in this group receive a dose-matched educational intervention with 12 visits by well-trained research therapists through face-to-face talks. Sessions focus on instruction on general information regarding stroke and rehabilitation, and a summary of participants' condition and progression is provided for each visit.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Strategy training for physical activity — STPA is a home-based rehabilitation that guides stroke participants to implement strategy training for addressing barriers to physical activity engagements. Participants learn and practice meta-cognitive strategies (to set a goal, to make a plan, to do the plan, to check the performance of the plan) throughout the intervention period.
  Other Names: STPA
  Arms: Strategy training for physical activity
Behavioral: Physical activity — PA program consists of a warm-up for 5 minutes, an aerobic exercise program for 30-40 minutes, a multicomponent exercise program (resistance and balance training) for 10-20 minutes, and finally, a cooling down program for 5 minutes.
  Other Names: PA
  Arms: Physical activity
Other: Education — Stroke-related information and knowledge that includes stroke subtypes and their etiology, risk factors of primary and secondary stroke, healthy lifestyles, common sequala, and adaptive skills for impaired functions are provided.
  Arms: Education

SUMMARY:
The goal of this randomized controlled trial is to examine if combining strategy training and physical activity (STPA) works to improve executive function in community-dwelling adults with post-stroke cognitive impairment. The main questions it aims to answer are:

* Does STPA and physical exercise alone lead to greater improvements in executive function among stroke survivors relative to the control intervention with education?
* Does STPA outperform physical exercise alone in the efficacy of executive functions?
* Do the effects of STPA on executive functions transfer to the global cognition, balance, and activity-participation outcomes?
* Do the effects of STPA persist for at least 6 months post-intervention?

Researchers will compare the efficacy of the STPA intervention against physical exercise alone or control intervention with education.

Participants will:

receive STPA, physical activity only, or an education program 2 to 3 sessions per week until finishing 12 sessions.

be assessed clinical outcomes at 5 times: pre-intervention, post-intervention, 3-month, 6-month, and 12-month follow-up.

DETAILED DESCRIPTION:
Poststroke cognitive impairment is a prevalent consequence of stroke that significantly impacts multifaceted outcomes. Executive functions are particularly responsive to training among cognitive domains. Despite the accumulating literature supporting physical activity interventions, their effects have been observed to be small and time-limited. Incorporating a behavioral approach, such as strategy training, offers a promising avenue for promoting improvements in executive functions and related stroke outcomes. To the best of investigators' understanding, no study has examined whether combining strategy training with physical activity-oriented goals can ameliorate executive and cognitive functions in individuals with stroke.

This study aims to examine and compare the efficacy of STPA and physical activity alone on executive, cognitive, activity, and participation functions in people with poststroke cognitive impairments. This study addresses the following specific aims:

1. Determine whether STPA in stroke patients with PSCI produces immediate improvements in executive functions that may generalize to improved global cognition, activity, or participation outcomes to a greater extent than a control intervention focused on stroke-related education;
2. Examine the potential association between improvements in executive functions resulting from STPA and enhancements in activity and participation performance;
3. Investigate the duration of therapeutic effects of STPA following the intervention;

To achieve these aims, a three-armed, parallel-design, randomized phase II clinical trial is designed and conducted. The investigators plan to recruit an expected sample of 120 adults with poststroke cognitive impairments from collaborative sites in northern Taiwan. Eligible participants are randomly assigned to one of the three intervention groups (STPA, physical activity, and education) at a 1:1:1 ratio. All participants should receive 12 sessions lasting 60 minutes over a maximum of 6 weeks. Primary outcomes for executive functions (Trail Making Test Part B and color-word condition of Stroop Color and Word Test) and secondary outcome measures, including Montreal Cognitive Assessment, processing speed (Trail Making Test Part A and word condition of Stroop Color and Word Test), Self-Regulation Skills Interview, Activity Measure for Post-Acute Care Outpatient Short Forms, Participation Measure-3 Domains, 4 Dimensions, Timed-Up and Go test, and Taiwan version of the International Physical Activity Questionnaire are administered at baseline (T1), post-intervention (T2), and 3-month (T3), 6-month (T4), and 12-month (T5) follow-ups. Data will be analyzed using constrained longitudinal data analysis and mixed-effects regression models. Additionally, qualitative in-depth interviews will be conducted with participants, caregivers, and therapists to understand their experiences, satisfaction, and their perceived effectiveness of the intervention. Transcribed data will be coded and analyzed with thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* A diagnosis of stroke within the past 3 year
* Speaking Mandarin
* Montreal Cognitive Assessment (maximum=30) < 26
* 14 item-Executive Interview > 3
* Willing to provide informed consent

Exclusion Criteria:

* Modified Rankin Scale (mRS) = 5
* Any conditions that may impede the participation in the study, such as severe aphasia, postoperative immobilization, or major neuropsychiatric diseases.
* Pre-stroke mRS >1
* 6-level Saltin-Grimby Physical Activity Level Scale (SGPALS) = 5 or 6
* Participating in other interventional study concurrently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Trail-Making Test, Part B (TMT-B) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  The TMT-B is a time-limited test (maximum 300 seconds) requiring participant to orderly trace stimuli that alternated between encircles numbers and characters as quickly and accurately as possible, with shorter time denoting better cognitive flexibility.
Stroop Color and Word Test, color-word condition (SCWT-CW) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  The Stroop Color and Word Test involves counting correct numbers according to a rule. In color-word condition, the word (e.g. "Red") is printed in a different color ink (e.g. green ink), while participants will require to name the color of ink, with greater correct responses denoting better inhibition.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  MoCA with 30 items evaluates the cognitive functions (range 0 to 30). This assessment covers domains such as visuospatial/executive skills, naming, memory, attention, language, abstraction, delayed recall, and orientation.
Trail-Making Test, Part A (TMT-A) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  The TMT-A requires participant to orderly trace the numeral stimuli as quickly and accurately as possible, and shorter time to complete represent better performance (maximum 300 seconds)
Stroop Color and Word Test, color condition (SCWT-C) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  The SCET-C asks participant to correctly answer the color ink in accordance with word on the cards, and greater correct responses denoting better performance.
Self-Regulation Skills Interview | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  This assessment comprises six standardized questions indicating three factors: awareness, readiness to change, and strategy behavior.
Activity Measure for Post-Acute Care (AM-PAC) Outpatient Short Forms | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  The AM-PAC measures the difficulty is performing three activity domains: Basic Mobility (18 activities), Daily Activity (15 activities), and Applied Cognition (19 activities) on a 4-point scale. In this trial, Applied Cognition domain is viewed as a secondary outcome.
Participation Measure-3 Domains, 4 Dimensions (PM-3D4D) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  PM-3D4D consists of 24 items for evaluating three domains of participation, which are community, productivity, and social. Participants will be asked to rate all items on the four distinct dimensions: (1) diversity, (2) frequency, (3) desire for change, and (4) perceived difficulty.
Time-Up and Go test (TUG) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  During the test, participants are asked to complete a serous of tasks: standing up from a chair, walking straight for 3 meters, turning around, walking back to the chair, and sitting down. The time to complete is recorded.
International Physical Activity Questionnaire (IPAQ) short form | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  IPAQ is used to calculate MET-minute per week based on participants' self-report physical activity durations on walking, moderate exercise, and vigorous exercise in the nearest 7 days.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  NIHSS is used to assess participants' stroke severity during the study period (range 0 to 42).
modified Rankin Scale (mRS) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  mRS is used to indicate participants' global disability during the study period (range 0 to 6).
Fugl-Meyer Assessment (FMA) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  FMA is used to quantify participants' motor impairment of upper and lower limb during the study period (range 0 to 100).
Saltin-Grimby Physical Activity Level Scale (SGPALS) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  SGPALS is used to indicate participants' level of physical activity during the study period (range 1 to 6).
Stroke Self-Efficacy Questionnaire (SSEQ) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  SSEQ is used to evaluate participants' self-efficacy during the study period.
EQ-5D-3L | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  EQ-5D-3L is used to evaluate participants' health-related quality of life during the study period.
Hospital Anxiety and Depression Scale (HADS) | 5 time points: baseline (T1), from baseline to the end of intervention at 5-6 weeks (T2), from the end of intervention to 3-month(T3), to 6-month (T4), and to 12-month follow-up (T5)
  HADS is used to measure participants' mood status during the study.

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Taipei Tzu Chi Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei